CLINICAL TRIAL: NCT03845075
Title: A 24-week Phase 2, Double-blind, Randomized, Placebo- Controlled, Single-center Safety and Efficacy Study to Evaluate Overall Safety and Tolerability of Co-administration of Tesofensine and Metoprolol in Subjects With Hypothalamic Injury-induced Obesity (HIO), and With a 24-week Open-label Extension, in Total 48 Weeks
Brief Title: 48 Weeks, Study to Evaluate Overall Safety and Tolerability of Co-administration of Tesofensine and Metoprolol in Subjects With Hypothalamic Injury-induced Obesity (HIO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TM005
Record Dates: First submitted 2019-01-30; First posted 2019-02-19 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hypothalamic Injury-induced Obesity (HIO)
MeSH Terms: interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active arm (Experimental): The active medication arm will be given co-administration of 0.5 mg tesofensine/50 mg metoprolol daily for 24 weeks.
  Interventions: Drug: Tesofensine/Metoprolol
- placebo arm (Placebo Comparator): The placebo arm will receive matching placebo tesofensine and placebo metoprolol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tesofensine/Metoprolol — During Part 1 subjects will be randomized to treatment with co-administration of 0.5 mg tesofensine/50mg metoprolol (active medication)
  Arms: active arm
Drug: Placebo — During Part 1 subjects will be randomized to matching placebo tesofensine and placebo metoprolol
  Arms: placebo arm

SUMMARY:
Double-blind, randomized, placebo-controlled, single- center study followed by an open-label extension period.

• The study will have two parts:

* Part 1: 24 weeks double-blind treatment (DB), followed by
* Part 2: 24 weeks open-label extension (OLE) - all subjects still participating at the end of Part 1 will be given an option to continue for additional 24 weeks on the active drug if evaluated eligible by the Investigator

DETAILED DESCRIPTION:
Part 1 - the double-blind (DB) part: The active medication arm will be given co-administration of 0.5 mg tesofensine/50 mg metoprolol daily for 24 weeks. The placebo arm will receive matching placebo tablets.

Part 2 - the open-label extension (OLE) part: All active participants at the end of the double-blind part will be given the active medication 0.5 mg tesofensine/50 mg metoprolol daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Males and females, aged 18-75
* Confirmed diagnosis of HIO
* BMI ≥27 kg/m2 (where overweight is related to the HIO)

Exclusion Criteria:

* Blood Pressure (BP) ≥160/90 mmHg
* Heart rate (HR) ≥ 90, <50 bpm
* Type 1 diabetes, Cushings disease, acromegaly, hypophysitis, infiltrative diseases or Prader-Willi syndrome
* Heart failure New York Heart Association (NYHA) level II or greater, decompensated heart failure
* Previous myocardial infarction or stroke within the last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD, DMSc, Principal Investigator — Department of Medical Endocrinology and metabolism Rigshospitalet,Copenhagen, DK
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 35 subjects with HIO were screened; 13 subjects were screen failures. A total of 21 unique subjects were assigned 22 randomization numbers. One subject was a screen failure who was randomized in error, and withdrawn after receiving 1 dose of tesofensine/metoprolol; this subject was later rescreened and rerandomized to placebo. This subject is summarized for both tesofensine/metoprolol and placebo (ie, considered as 2 independent subjects).
Groups:
- Tesofensine/Metoprolol: Subjects were randomized to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol (active medication) once daily for 24 weeks during Part 1.
- Placebo: Subjects were randomized to receive matching placebo tesofensine and placebo metoprolol once daily for 24 weeks during Part 1.
- Tesofensine/Metoprolol -> Tesofensine/Metoprolol: Subjects who received co-administration of 0.5 mg tesofensine/50 mg metoprolol (active medication) once daily for 24 weeks during Part 1 and continued to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol once daily for an additional 24 weeks in Part 2.
- Placebo -> Tesofensine/Metoprolol: Subjects who received matching placebo tesofensine and placebo metoprolol once daily for 24 weeks during Part 1 and were switched to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol once daily for an additional 24 weeks in Part 2.
Period: Part 1 - DB
Arm/Group | Tesofensine/Metoprolol | Placebo | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Started | 14 | 8 | 0 | 0
Completed | 12 | 6 | 0 | 0
Not Completed | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Screen failure, but received 1 dose of study drug in error | 1 | 0 | 0 | 0
Period: Part 2 - OLE
Arm/Group | Tesofensine/Metoprolol | Placebo | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Started | 0 | 0 | 12 | 6
Completed | 0 | 0 | 12 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects were randomized to receive matching placebo tablets once daily for 24 weeks during Part 1.
- Total: Total of all reporting groups
Arm/Group | Tesofensine/Metoprolol | Placebo | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.3) | 44.4 (18.3) | 45.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 14 | 8 | 22
Weight [Mean (Standard Deviation); unit: kg] | 114.34 (18.14) | 112.16 (27.04) | 113.55 (21.18)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number and percentage of participants with adverse events in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: Safety Analysis Set: all subjects who took at least one dose of the IMPs (active substances or placebos)
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants | 12 | 7

2. Primary Outcome: Number of Participants With at Least One Mild, Moderate or Severe Adverse Event
Description: Number and percentage of participants with mild, moderate or severe adverse events in each of the two treatment arms.
Time Frame: from Baseline to week 24
Population: Safety Analysis Set: all subjects who took at least one dose of the IMPs (active substances or placebos)
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  At least one mild AE | 11 | 7
  At least one moderate AE | 10 | 5
  At least one severe AE | 2 | 2

3. Primary Outcome: Participants (Number and Percentage) With and Type of Serious Adverse Events
Description: Number and percentage of participants with at least one serious adverse event, indicating type, in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: Safety Analysis Set: all subjects who took at least one dose of the IMPs (active substances or placebos)
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  At least one SAE | 2 | 1
  Preferred Term: Anxiety | 1 | 0
  Preferred Term: Craniopharyngioma | 1 | 0
  Preferred Term: Hyponatraemia | 0 | 1
  Preferred Term: Post procedural complication | 1 | 0

4. Primary Outcome: Safety as Assessed by Systolic Blood Pressure [mmHg]
Description: Systolic blood pressure in mmHg measured at each visit in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: Safety Analysis Set: all subjects who took at least one dose of the IMPs (active substances or placebos). Subjects with an assessment at given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 13 | 8
mmHg
  Baseline | 124.0 (9) | 134.5 (16)
  Week 4 | 126.6 (12) | 131.8 (17)
  Week 8: number analyzed (Participants) | 12 | 6
  Week 8 | 129.2 (17) | 126.3 (23)
  Week 12: number analyzed (Participants) | 12 | 6
  Week 12 | 126.3 (13) | 126.2 (14)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 123.9 (14) | 126.0 (17)
  Week 20: number analyzed (Participants) | 12 | 6
  Week 20 | 127.3 (12) | 129.2 (18)
  Week 24: number analyzed (Participants) | 12 | 6
  Week 24 | 125.3 (16) | 130.5 (22)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; Week 4; Safety set; LOCF; Test type: Superiority; p = 0.4671, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 3.60, 95% CI 2-sided [-6.58 to 13.78] — Estimate and 95% CI are based on a least squares (LS) mean difference from an ANCOVA model with treatment as factor and baseline as covariate
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol vs Placebo; Week 8; Safety set; LOCF; Test type: Superiority; p = 0.1808, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 10.11, 95% CI 2-sided [-5.14 to 25.36] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol vs Placebo; Week 12; Safety set; LOCF; Test type: Superiority; p = 0.4171, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 4.63, 95% CI 2-sided [-7.08 to 16.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol vs Placebo; Week 16; Safety set; LOCF; Test type: Superiority; p = 0.3116, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 5.33, 95% CI 2-sided [-5.43 to 16.10] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol vs Placebo; Week 20; Safety set; LOCF; Test type: Superiority; p = 0.2353, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 5.80, 95% CI 2-sided [-4.12 to 15.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol vs Placebo; Week 24; Safety set; LOCF; Test type: Superiority; p = 0.3037, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 5.86, 95% CI 2-sided [-5.76 to 17.48] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Safety as Assessed by Diastolic Blood Pressure [mmHg]
Description: Diastolic blood pressure in mmHg measured at each visit in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 13 | 8
mmHg
  Baseline | 83.2 (14) | 85.9 (8)
  Week 4 | 84.2 (8) | 86.8 (8)
  Week 8: number analyzed (Participants) | 12 | 6
  Week 8 | 84.5 (9) | 86.0 (9)
  Week 12: number analyzed (Participants) | 12 | 6
  Week 12 | 81.5 (10) | 86.5 (8)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 81.4 (9) | 80.3 (13)
  Week 20: number analyzed (Participants) | 12 | 6
  Week 20 | 84.3 (9) | 85.7 (9)
  Week 24: number analyzed (Participants) | 12 | 6
  Week 24 | 83.1 (9) | 84.2 (13)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; Week 4; Safety set; LOCF; Test type: Superiority; p = 0.6543, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.31, 95% CI 2-sided [-7.33 to 4.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol vs Placebo; Week 8; Safety set; LOCF; Test type: Superiority; p = 0.7941, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.94, 95% CI 2-sided [-6.50 to 8.38] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol vs Placebo; Week 12; Safety set; LOCF; Test type: Superiority; p = 0.5937, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.00, 95% CI 2-sided [-9.72 to 5.73] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol vs Placebo; Week 16; Safety set; LOCF; Test type: Superiority; p = 0.5423, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.56, 95% CI 2-sided [-6.11 to 11.23] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol vs Placebo; Week 20; Safety set; LOCF; Test type: Superiority; p = 0.7226, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.20, 95% CI 2-sided [-5.77 to 8.16] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol vs Placebo; Week 24; Safety set; LOCF; Test type: Superiority; p = 0.7912, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.15, 95% CI 2-sided [-7.85 to 10.16] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Safety as Assessed by Heart Rate [Bpm]
Description: Heart rate measured in beats per minute (bpm) at each visit in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 13 | 8
bpm
  Baseline | 75.5 (8) | 78.9 (11)
  Week 4 | 71.9 (9) | 75.9 (12)
  Week 8: number analyzed (Participants) | 12 | 6
  Week 8 | 72.7 (8) | 76.0 (13)
  Week 12: number analyzed (Participants) | 12 | 6
  Week 12 | 74.2 (10) | 73.3 (8)
  Week 16: number analyzed (Participants) | 12 | 6
  Week 16 | 73.8 (13) | 74.8 (6)
  Week 20: number analyzed (Participants) | 12 | 6
  Week 20 | 74.8 (11) | 77.2 (13)
  Week 24: number analyzed (Participants) | 12 | 6
  Week 24 | 73.6 (10) | 71.5 (9)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; Week 4; Safety set; LOCF; Test type: Superiority; p = 0.7023, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.35, 95% CI 2-sided [-8.67 to 5.97] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol vs Placebo; Week 8; Safety set; LOCF; Test type: Superiority; p = 0.9012, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.48, 95% CI 2-sided [-8.58 to 7.61] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol vs Placebo; Week 12; Safety set; LOCF; Test type: Superiority; p = 0.6138, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.14, 95% CI 2-sided [-6.63 to 10.92] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol vs Placebo; Week 16; Safety set; LOCF; Test type: Superiority; p = 0.7889, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.23, 95% CI 2-sided [-8.26 to 10.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol vs Placebo; Week 20; Safety set; LOCF; Test type: Superiority; p = 0.9536, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.30, 95% CI 2-sided [-10.34 to 10.94] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol vs Placebo; Week 24; Safety set; LOCF; Test type: Superiority; p = 0.5551, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.70, 95% CI 2-sided [-6.72 to 12.12] — [estimate comment as in outcome 4, analysis 1]

7. Primary Outcome: Safety as Assessed by Hematology Parameters
Description: Number and percentage of deviations from normal range (as defined by the investigational site's laboratory) for hemoglobin, platelet counts, white cells count, differential counts at baseline, week 12 and week 24 in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  Hemoglobin: Baseline - Low | 0 | 0
  Hemoglobin: Baseline - High | 0 | 1
  Hemoglobin: Week 12 - Low: number analyzed (Participants) | 13 | 8
  Hemoglobin: Week 12 - Low | 0 | 0
  Hemoglobin: Week 12 - High: number analyzed (Participants) | 13 | 8
  Hemoglobin: Week 12 - High | 0 | 0
  Hemoglobin: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Hemoglobin: Week 24 - Low | 1 | 0
  Hemoglobin: Week 24 - High: number analyzed (Participants) | 12 | 6
  Hemoglobin: Week 24 - High | 0 | 0
  Platelets: Baseline - Low | 0 | 0
  Platelets: Baseline - High | 1 | 0
  Platelets: Week 12 - Low: number analyzed (Participants) | 13 | 8
  Platelets: Week 12 - Low | 0 | 0
  Platelets: Week 12 - High: number analyzed (Participants) | 13 | 8
  Platelets: Week 12 - High | 1 | 0
  Platelets: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Platelets: Week 24 - Low | 0 | 0
  Platelets: Week 24 - High: number analyzed (Participants) | 12 | 6
  Platelets: Week 24 - High | 1 | 0
  WBC: Baseline - Low | 0 | 0
  WBC: Baseline - High | 3 | 2
  WBC: Week 12 - Low: number analyzed (Participants) | 13 | 8
  WBC: Week 12 - Low | 0 | 0
  WBC: Week 12 - High: number analyzed (Participants) | 13 | 8
  WBC: Week 12 - High | 5 | 1
  WBC: Week 24 - Low: number analyzed (Participants) | 12 | 6
  WBC: Week 24 - Low | 0 | 0
  WBC: Week 24 - High: number analyzed (Participants) | 12 | 6
  WBC: Week 24 - High | 0 | 1
  Neutrophils: Baseline - Low | 1 | 0
  Neutrophils: Baseline - High | 1 | 1
  Neutrophils: Week 12 - Low: number analyzed (Participants) | 13 | 8
  Neutrophils: Week 12 - Low | 0 | 0
  Neutrophils: Week 12 - High: number analyzed (Participants) | 13 | 8
  Neutrophils: Week 12 - High | 4 | 1
  Neutrophils: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Neutrophils: Week 24 - Low | 1 | 0
  Neutrophils: Week 24 - High: number analyzed (Participants) | 12 | 6
  Neutrophils: Week 24 - High | 1 | 1
  Monocytes: Baseline - Low | 0 | 0
  Monocytes: Baseline - High | 0 | 0
  Monocytes: Week 12 - Low: number analyzed (Participants) | 13 | 8
  Monocytes: Week 12 - Low | 0 | 0
  Monocytes: Week 12 - High: number analyzed (Participants) | 13 | 8
  Monocytes: Week 12 - High | 1 | 0
  Monocytes: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Monocytes: Week 24 - Low | 0 | 0
  Monocytes: Week 24 - High: number analyzed (Participants) | 12 | 6
  Monocytes: Week 24 - High | 1 | 0
  Lymphocytes: Baseline - Low | 0 | 1
  Lymphocytes: Baseline - High | 1 | 2
  Lymphocytes: Week 12 - Low: number analyzed (Participants) | 13 | 8
  Lymphocytes: Week 12 - Low | 0 | 1
  Lymphocytes: Week 12 - High: number analyzed (Participants) | 13 | 8
  Lymphocytes: Week 12 - High | 0 | 0
  Lymphocytes: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Lymphocytes: Week 24 - Low | 0 | 0
  Lymphocytes: Week 24 - High: number analyzed (Participants) | 12 | 6
  Lymphocytes: Week 24 - High | 1 | 0

8. Primary Outcome: Safety as Assessed by Electrolytes and Creatinine
Description: Number and percentage of deviations from normal range (as defined by the investigational site's laboratory) for sodium, potassium, creatinine at each visit in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  Sodium: Baseline - Low | 0 | 0
  Sodium: Baseline - High | 2 | 2
  Sodium: Week 4 - Low: number analyzed (Participants) | 13 | 8
  Sodium: Week 4 - Low | 0 | 0
  Sodium: Week 4 - High: number analyzed (Participants) | 13 | 8
  Sodium: Week 4 - High | 0 | 0
  Sodium: Week 8 - Low: number analyzed (Participants) | 13 | 7
  Sodium: Week 8 - Low | 0 | 0
  Sodium: Week 8 - High: number analyzed (Participants) | 13 | 7
  Sodium: Week 8 - High | 1 | 1
  Sodium: Week 12 - Low: number analyzed (Participants) | 12 | 6
  Sodium: Week 12 - Low | 0 | 0
  Sodium: Week 12 - High: number analyzed (Participants) | 12 | 6
  Sodium: Week 12 - High | 1 | 0
  Sodium: Week 16 - Low: number analyzed (Participants) | 12 | 6
  Sodium: Week 16 - Low | 0 | 0
  Sodium: Week 16 - High: number analyzed (Participants) | 12 | 6
  Sodium: Week 16 - High | 1 | 0
  Sodium: Week 20 - Low: number analyzed (Participants) | 12 | 6
  Sodium: Week 20 - Low | 0 | 0
  Sodium: Week 20 - High: number analyzed (Participants) | 12 | 6
  Sodium: Week 20 - High | 2 | 2
  Sodium: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Sodium: Week 24 - Low | 1 | 0
  Sodium: Week 24 - High: number analyzed (Participants) | 12 | 6
  Sodium: Week 24 - High | 0 | 1
  Potassium: Baseline - Low | 0 | 0
  Potassium: Baseline - High | 0 | 1
  Potassium: Week 4 - Low: number analyzed (Participants) | 13 | 8
  Potassium: Week 4 - Low | 2 | 1
  Potassium: Week 4 - High: number analyzed (Participants) | 13 | 8
  Potassium: Week 4 - High | 0 | 1
  Potassium: Week 8 - Low: number analyzed (Participants) | 13 | 7
  Potassium: Week 8 - Low | 2 | 0
  Potassium: Week 8 - High: number analyzed (Participants) | 13 | 7
  Potassium: Week 8 - High | 0 | 0
  Potassium: Week 12 - Low: number analyzed (Participants) | 12 | 6
  Potassium: Week 12 - Low | 1 | 0
  Potassium: Week 12 - High: number analyzed (Participants) | 12 | 6
  Potassium: Week 12 - High | 0 | 0
  Potassium: Week 16 - Low: number analyzed (Participants) | 12 | 6
  Potassium: Week 16 - Low | 1 | 0
  Potassium: Week 16 - High: number analyzed (Participants) | 12 | 6
  Potassium: Week 16 - High | 0 | 1
  Potassium: Week 20 - Low: number analyzed (Participants) | 12 | 6
  Potassium: Week 20 - Low | 1 | 0
  Potassium: Week 20 - High: number analyzed (Participants) | 12 | 6
  Potassium: Week 20 - High | 0 | 0
  Potassium: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Potassium: Week 24 - Low | 0 | 1
  Potassium: Week 24 - High: number analyzed (Participants) | 12 | 6
  Potassium: Week 24 - High | 0 | 0
  Creatinine: Baseline - Low | 3 | 2
  Creatinine: Baseline - High | 0 | 0
  Creatinine: Week 4 - Low: number analyzed (Participants) | 13 | 8
  Creatinine: Week 4 - Low | 2 | 4
  Creatinine: Week 4 - High: number analyzed (Participants) | 13 | 8
  Creatinine: Week 4 - High | 0 | 0
  Creatinine: Week 8 - Low: number analyzed (Participants) | 13 | 7
  Creatinine: Week 8 - Low | 2 | 3
  Creatinine: Week 8 - High: number analyzed (Participants) | 13 | 7
  Creatinine: Week 8 - High | 0 | 0
  Creatinine: Week 12 - Low: number analyzed (Participants) | 12 | 6
  Creatinine: Week 12 - Low | 2 | 2
  Creatinine: Week 12 - High: number analyzed (Participants) | 12 | 6
  Creatinine: Week 12 - High | 0 | 0
  Creatinine: Week 16 - Low: number analyzed (Participants) | 12 | 6
  Creatinine: Week 16 - Low | 3 | 2
  Creatinine: Week 16 - High: number analyzed (Participants) | 12 | 6
  Creatinine: Week 16 - High | 0 | 0
  Creatinine: Week 20 - Low: number analyzed (Participants) | 12 | 6
  Creatinine: Week 20 - Low | 4 | 2
  Creatinine: Week 20 - High: number analyzed (Participants) | 12 | 6
  Creatinine: Week 20 - High | 0 | 0
  Creatinine: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Creatinine: Week 24 - Low | 3 | 1
  Creatinine: Week 24 - High: number analyzed (Participants) | 12 | 6
  Creatinine: Week 24 - High | 0 | 0

9. Primary Outcome: Safety as Assessed by Liver and Kidney Function Tests
Description: Number and percentage of deviations from normal range (as defined by the investigational site's laboratory) for gamma glutamyl transferase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), glomerular filtration rate (GFR), and urea at baseline, week 12, and week 24 in each of the two treatment arms
Time Frame: from Baseline to week 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  GGT: Baseline - Low | 0 | 0
  GGT: Baseline - High | 5 | 1
  GGT: Week 12 - Low: number analyzed (Participants) | 13 | 8
  GGT: Week 12 - Low | 0 | 1
  GGT: Week 12 - High: number analyzed (Participants) | 13 | 8
  GGT: Week 12 - High | 5 | 2
  GGT: Week 24 - Low: number analyzed (Participants) | 12 | 6
  GGT: Week 24 - Low | 0 | 0
  GGT: Week 24 - High: number analyzed (Participants) | 12 | 6
  GGT: Week 24 - High | 4 | 0
  AST: Baseline - Low | 0 | 0
  AST: Baseline - High | 0 | 0
  AST: Week 12 - Low: number analyzed (Participants) | 12 | 8
  AST: Week 12 - Low | 0 | 0
  AST: Week 12 - High: number analyzed (Participants) | 12 | 8
  AST: Week 12 - High | 0 | 0
  AST: Week 24 - Low: number analyzed (Participants) | 12 | 6
  AST: Week 24 - Low | 0 | 0
  AST: Week 24 - High: number analyzed (Participants) | 12 | 6
  AST: Week 24 - High | 0 | 0
  ALT: Baseline - Low | 0 | 0
  ALT: Baseline - High | 0 | 0
  ALT: Week 12 - Low: number analyzed (Participants) | 13 | 8
  ALT: Week 12 - Low | 0 | 0
  ALT: Week 12 - High: number analyzed (Participants) | 13 | 8
  ALT: Week 12 - High | 1 | 0
  ALT: Week 24 - Low: number analyzed (Participants) | 12 | 6
  ALT: Week 24 - Low | 0 | 0
  ALT: Week 24 - High: number analyzed (Participants) | 12 | 6
  ALT: Week 24 - High | 0 | 0
  ALP: Baseline - Low | 0 | 0
  ALP: Baseline - High | 1 | 0
  ALP: Week 12 - Low: number analyzed (Participants) | 13 | 8
  ALP: Week 12 - Low | 0 | 0
  ALP: Week 12 - High: number analyzed (Participants) | 13 | 8
  ALP: Week 12 - High | 2 | 0
  ALP: Week 24 - Low: number analyzed (Participants) | 12 | 6
  ALP: Week 24 - Low | 0 | 0
  ALP: Week 24 - High: number analyzed (Participants) | 12 | 6
  ALP: Week 24 - High | 1 | 0
  GFR: Baseline - Low: number analyzed (Participants) | 12 | 8
  GFR: Baseline - Low | 0 | 0
  GFR: Baseline - High: number analyzed (Participants) | 12 | 8
  GFR: Baseline - High | 0 | 0
  GFR: Week 12 - Low: number analyzed (Participants) | 12 | 7
  GFR: Week 12 - Low | 0 | 0
  GFR: Week 12 - High: number analyzed (Participants) | 12 | 7
  GFR: Week 12 - High | 0 | 0
  GFR: Week 24 - Low: number analyzed (Participants) | 11 | 6
  GFR: Week 24 - Low | 0 | 0
  GFR: Week 24 - High: number analyzed (Participants) | 11 | 6
  GFR: Week 24 - High | 0 | 0
  Urea: Baseline - Low: number analyzed (Participants) | 14 | 7
  Urea: Baseline - Low | 1 | 1
  Urea: Baseline - High: number analyzed (Participants) | 14 | 7
  Urea: Baseline - High | 0 | 0
  Urea: Week 12 - Low: number analyzed (Participants) | 11 | 5
  Urea: Week 12 - Low | 2 | 0
  Urea: Week 12 - High: number analyzed (Participants) | 11 | 5
  Urea: Week 12 - High | 0 | 0
  Urea: Week 24 - Low: number analyzed (Participants) | 12 | 6
  Urea: Week 24 - Low | 1 | 0
  Urea: Week 24 - High: number analyzed (Participants) | 12 | 6
  Urea: Week 24 - High | 0 | 0

10. Secondary Outcome: Composite Satiety Score (CSS)
Description: Change in satiety and appetite using the CSS from Baseline to week 24, from Baseline to week 48 and from week 24 to week 48 measured at each visit for each of the two treatment arms
  Full name of the scale: composite satiety score (CSS), sometimes referred to as "appetite suppression score". Range of values is 0-100; lower the value, hungrier a person is. CSS = (satiety + fullness + [100 - hunger] + [100 - prospective food consumption]) / 4. The four variables included are measured by visual analog scales (0-100 mm)
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: Modified Intention-to-treat (mITT) Population: all subjects who entered Part 2 (open-label extension) and had nonmissing baseline assessments and at least 1 post-Part 1 assessment. Last observation carried forward (LOCF) approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tesofensine/Metoprolol -> Tesofensine/Metoprolol: Subjects who received co-administration of 0.5 mg tesofensine/50 mg metoprolol (active medication) once daily for 24 weeks during Part 1 continued to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol once daily for an additional 24 weeks in Part 2.
- Placebo -> Tesofensine/Metoprolol: Subjects who received matching placebo tablets once daily for 24 weeks during Part 1 were switched to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol once daily for an additional 24 weeks in Part 2.
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
score on a scale
  Baseline to Week 24 | 4.5 (20.6) | 6.5 (19.3)
  Baseline to Week 48 | 4.2 (15.1) | 11.2 (14.3)
  Week 24 to Week 48 | -0.3 (14.4) | 4.7 (12.5)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; Test type: Superiority; p = 0.7782, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.52, 95% CI 2-sided [-21.23 to 16.20] — (Tesofensine/Metoprolol -> Tesofensine/Metoprolol) - (Placebo -> Tesofensine/Metoprolol). Estimate and 95% CI are based on a least squares (LS) mean difference from an ANCOVA model with treatment as factor and baseline as covariate
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; Test type: Superiority; p = 0.3130, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -7.26, 95% CI 2-sided [-22.09 to 7.56] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to Week 48; Test type: Superiority; p = 0.4033, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -5.73, 95% CI 2-sided [-19.92 to 8.47] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Body Weight
Description: Change in body weight from baseline to week 24, from baseline to 48 and from week 24 to week 48 measured at each visit for each of the two treatment arms
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
kg
  Baseline to Week 24 | -7.93 (6.59) | -0.15 (4.74)
  Baseline to Week 48 | -6.53 (7.36) | -5.65 (8.90)
  Week 24 to Week 48 | 1.40 (4.05) | -5.50 (6.20)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; Test type: Superiority; p = 0.0325, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -7.50, 95% CI 2-sided [-14.29 to -0.71] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; Test type: Superiority; p = 0.9394, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.32, 95% CI 2-sided [-9.04 to 8.40] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol; Week 24 to Week 28; Test type: Superiority; p = 0.0135, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 6.91, 95% CI 2-sided [1.65 to 12.18] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Body Composition - Fat Mass
Description: Change in body fat mass as measured in kg by DXA scan measured at baseline, week 24 and week 48 for each of the two treatment arms. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: Modified Intention-to-treat (mITT) Population: all subjects who entered Part 2 (open-label extension) and had nonmissing baseline assessments and at least 1 post-Part 1 assessment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
kg
  Baseline to Week 24 | -5.31 (5.34) | -1.04 (3.75)
  Baseline to Week 48 | -4.87 (5.31) | -3.77 (5.81)
  Week 24 to Week 48 | 0.44 (3.50) | -2.73 (3.37)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed; Test type: Superiority; p = 0.1048, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -4.17, 95% CI 2-sided [-9.31 to 0.98] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT observed; Test type: Superiority; p = 0.7189, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.99, 95% CI 2-sided [-6.75 to 4.77] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to Week 48; mITT observed; Test type: Superiority; p = 0.1053, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 3.09, 95% CI 2-sided [-0.73 to 6.91] — [estimate comment as in outcome 10, analysis 1]

13. Secondary Outcome: Body Composition - Lean Body Mass
Description: Change in lean body mass as measured in kg by DXA scan measured at baseline, week 24 and week 48 for each of the two treatment arms. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
kg
  Baseline to Week 24 | -2.85 (1.88) | 0.55 (1.32)
  Baseline to Week 48 | -1.81 (2.18) | -1.87 (3.36)
  Week 24 to Week 48 | 1.04 (1.18) | -2.42 (3.51)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed; Test type: Superiority; p = 0.0033, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -3.12, 95% CI 2-sided [-5.02 to -1.21] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF; Test type: Superiority; p = 0.6663, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.58, 95% CI 2-sided [-2.24 to 3.41] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to Week 48; mITT LOCF; Test type: Superiority; p = 0.0058, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 3.59, 95% CI 2-sided [1.21 to 5.98] — [estimate comment as in outcome 10, analysis 1]

14. Secondary Outcome: Glycemic Control - HbA1c
Description: Change in HbA1c from baseline to week 24, baseline to week 48 and week 24 to week 48 for each of the two treatment arms. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
mmol/mol
  Baseline to Week 24 | -6.00 (15.39) | -0.17 (2.40)
  Baseline to Week 48 | -5.33 (14.79) | -0.17 (2.23)
  Week 24 to Week 48 | 0.67 (1.30) | 0.00 (0.63)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed; Test type: Superiority; p = 0.0713, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -3.02, 95% CI 2-sided [-6.34 to 0.30] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF; Test type: Superiority; p = 0.1457, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.48, 95% CI 2-sided [-5.92 to 0.96] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to Week 48; mITT LOCF; Test type: Superiority; p = 0.1837, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.85, 95% CI 2-sided [-0.45 to 2.15] — [estimate comment as in outcome 10, analysis 1]

15. Secondary Outcome: Glycemic Control - Fasting Plasma Glucose
Description: Change in fasting plasma glucose from baseline to week 24, baseline to week 48 and week 24 to week 48 measured at each visit for each of the two treatments arms. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
mmol/L
  Baseline to Week 24 | -0.29 (0.64) | -0.28 (0.57)
  Baseline to Week 48 | -0.11 (0.53) | 0.08 (0.37)
  Week 24 to Week 48 | 0.18 (0.46) | 0.37 (0.59)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT LOCF; Test type: Superiority; p = 0.7926, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.05, 95% CI 2-sided [-0.42 to 0.33] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF; Test type: Superiority; p = 0.2124, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.27, 95% CI 2-sided [-0.72 to 0.17] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to Week 48; mITT LOCF; Test type: Superiority; p = 0.6084, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.14, 95% CI 2-sided [-0.72 to 0.43] — [estimate comment as in outcome 10, analysis 1]

16. Secondary Outcome: Craving for Something Sweet, Salty, Meat/Fish, or Fatty
Description: Change in craving for something sweet, salty, meat/fish, or fatty by the use of visual analogue scales (VAS) from baseline to week 24, from baseline to week 48, and from week 24 to week 48
  The VAS consisted of a 100-mm horizontal line; subjects placed a vertical line on the VAS to indicate the level of intensity of their food craving. The VAS value is the distance in mm (0-100 mm) from the left end of the line to the subject's vertical line (higher value represents less craving).
  mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
score on a scale
  Desire for something sweet from baseline to week 24 | 9.0 (36.6) | 16.2 (30.8)
  Desire for something sweet from baseline to week 48 | 2.1 (35.8) | 35.3 (32.9)
  Desire for something sweet from week 24 to week 48 | -6.9 (20.2) | 19.2 (30.7)
  Desire for something salty from baseline to week 24 | -2.3 (27.9) | 13.2 (21.5)
  Desire for something salty from baseline to week 48 | -3.4 (28.8) | 33.3 (30.9)
  Desire for something salty from week 24 to week 48 | -1.2 (8.5) | 20.2 (22.7)
  Desire for meat/fish from baseline to week 24 | 7.3 (42.6) | 8.8 (34.0)
  Desire for meat/fish from baseline to week 48 | 14.0 (44.1) | 35.0 (34.6)
  Desire for meat/fish from week 24 to week 48 | 6.8 (18.6) | 26.2 (34.2)
  Desire for something fatty from baseline to week 24 | 18.2 (22.6) | 2.2 (11.3)
  Desire for something fatty from baseline to week 48 | 5.2 (25.7) | 22.5 (26.3)
  Desire for something fatty from week 24 to week 48 | -13.0 (15.6) | 20.3 (28.0)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to week 24; mITT observed. (Like to eat something fatty); Test type: Superiority; p = 0.0905, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 16.00, 95% CI 2-sided [-2.85 to 34.85] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Like some meat/fish); Test type: Superiority; p = 0.6285, ANCOVA — P-value from ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 6.65, 95% CI 2-sided [-22.05 to 35.36] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Eat something salty); Test type: Superiority; p = 0.5884, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -6.81, 95% CI 2-sided [-33.05 to 19.43] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Eat something sweet); Test type: Superiority; p = 0.8533, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.98, 95% CI 2-sided [-30.73 to 36.68] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Like to eat something fatty); Test type: Superiority; p = 0.1529, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -17.33, 95% CI 2-sided [-41.87 to 7.20] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Like some meat/fish); Test type: Superiority; p = 0.3399, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -11.75, 95% CI 2-sided [-37.15 to 13.65] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 7: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Eat something salty); Test type: Superiority; p = 0.0673, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -23.95, 95% CI 2-sided [-49.84 to 1.93] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 8: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Eat something sweet); Test type: Superiority; p = 0.1657, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -22.60, 95% CI 2-sided [-55.65 to 10.46] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 9: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Like to eat something fatty); Test type: Superiority; p = 0.0108, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -30.18, 95% CI 2-sided [-52.31 to -8.06] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Like some meat/fish); Test type: Superiority; p = 0.1710, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -14.79, 95% CI 2-sided [-36.71 to 7.13] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Eat something salty); Test type: Superiority; p = 0.0083, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -19.86, 95% CI 2-sided [-33.80 to -5.93] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 12: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Eat something sweet); Test type: Superiority; p = 0.0631, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -22.98, 95% CI 2-sided [-47.39 to 1.43] — [estimate comment as in outcome 10, analysis 1]

17. Secondary Outcome: Thirst
Description: Change in thirst by the use of a visual analog scale (VAS) from baseline to week 24, from baseline to week 48, and from week 24 to week 48
  The VAS consisted of a 100-mm horizontal line; subjects placed a vertical line on the VAS to indicate the level of intensity of their thirst. The VAS value is the distance in mm (0-100 mm) from the left end of the line to the subject's vertical line (higher value represents an increase in perception of thirst).
  mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
score on a scale
  From baseline to week 24 | -2.4 (28.9) | -18.8 (23.2)
  From baseline to week 48 | -6.3 (25.8) | -16.7 (18.8)
  From week 24 to week 48 | -3.8 (16.5) | 2.2 (20.5)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed; Test type: Superiority; p = 0.8082, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.56, 95% CI 2-sided [-24.65 to 19.53] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF; Test type: Superiority; p = 0.9034, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.42, 95% CI 2-sided [-25.94 to 23.10] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF; Test type: Superiority; p = 0.4658, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -7.00, 95% CI 2-sided [-26.93 to 12.93] — [estimate comment as in outcome 10, analysis 1]

18. Secondary Outcome: Waist Circumference
Description: Change in waist circumference from baseline to week 24, from baseline to week 48, and from week 24 to week 48. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
cm
  From baseline to week 24 | -7.08 (6.93) | -1.17 (4.40)
  From baseline to week 48 | -5.75 (5.26) | -3.00 (6.51)
  From week 24 to week 48 | 1.33 (4.01) | -1.83 (2.64)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT LOCF; Test type: Superiority; p = 0.0537, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -5.68, 95% CI 2-sided [-11.46 to 0.10] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF; Test type: Superiority; p = 0.3772, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.69, 95% CI 2-sided [-8.98 to 3.61] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF; Test type: Superiority; p = 0.1171, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 3.03, 95% CI 2-sided [-0.85 to 6.91] — [estimate comment as in outcome 10, analysis 1]

19. Secondary Outcome: Lipid Profile
Description: Change in lipid profile from baseline to week 24, from baseline to week 48, and from week 24 to week 48. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
mmol/L
  Change in total cholesterol from baseline to week 24 | -0.17 (0.46) | -0.17 (0.45)
  Change in total cholesterol from baseline to week 48 | -0.01 (0.60) | -0.22 (0.75)
  Change in total cholesterol from week 24 to week 48 | 0.16 (0.48) | -0.05 (0.69)
  Change in HDL cholesterol from baseline to week 24 | 0.04 (0.21) | -0.02 (0.37)
  Change in HDL cholesterol from baseline to week 48 | 0.09 (0.26) | 0.03 (0.25)
  Change in HDL cholesterol from week 24 to week 48 | 0.05 (0.24) | 0.05 (0.16)
  Change in LDL cholesterol from baseline to week 24 | -0.23 (0.39) | -0.20 (0.43)
  Change in LDL cholesterol from baseline to week 48 | -0.15 (0.38) | -0.32 (0.53)
  Change in LDL cholesterol from week 24 to week 48 | 0.08 (0.28) | -0.12 (0.45)
  Change in triglycerides from baseline to week 24 | -0.08 (0.77) | -0.30 (0.76)
  Change in triglycerides from baseline to week 48 | -0.07 (0.77) | -0.48 (0.28)
  Change in triglycerides from week 24 to week 48 | 0.01 (0.69) | -0.18 (0.66)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Change in total cholesterol); Test type: Superiority; p = 0.8623, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.05, 95% CI 2-sided [-0.59 to 0.50] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Change in HDL cholesterol); Test type: Superiority; p = 0.8327, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.03, 95% CI 2-sided [-0.25 to 0.30] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Change in LDL cholesterol); Test type: Superiority; p = 0.8080, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.06, 95% CI 2-sided [-0.53 to 0.42] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 24; mITT observed. (Change in triglycerides); Test type: Superiority; p = 0.5791, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.62 to 1.07] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Change in cholesterol); Test type: Superiority; p = 0.9337, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.03, 95% CI 2-sided [-0.71 to 0.77] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Change in HDL cholesterol); Test type: Superiority; p = 0.9305, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.01, 95% CI 2-sided [-0.21 to 0.23] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 7: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Change in LDL cholesterol); Test type: Superiority; p = 0.6910, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.09, 95% CI 2-sided [-0.40 to 0.59] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 8: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Baseline to Week 48; mITT LOCF. (Change in triglycerides); Test type: Superiority; p = 0.2688, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.35, 95% CI 2-sided [-0.30 to 1.01] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 9: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Change in cholesterol); Test type: Superiority; p = 0.8262, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.06, 95% CI 2-sided [-0.54 to 0.67] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Change in HDL cholesterol); Test type: Superiority; p = 0.8293, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -0.02, 95% CI 2-sided [-0.20 to 0.17] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Change in LDL cholesterol); Test type: Superiority; p = 0.5486, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.11, 95% CI 2-sided [-0.27 to 0.49] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 12: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Change in triglycerides); Test type: Superiority; p = 0.3226, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.24, 95% CI 2-sided [-0.26 to 0.75] — [estimate comment as in outcome 10, analysis 1]

20. Secondary Outcome: Quality of Life - SF-36
Description: Change in quality of life by use of the Short Form 36 Health Survey (SF-36) scores from baseline to week 24, from baseline to week 48, and from week 24 to week 48
  The physical component summary score includes the aggregated scores for scales of physical functioning, role-physical, bodily pain, and general health. The mental health component summary score includes the aggregated scores for scales of vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100; higher score indicates better health.
  mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
score on a scale
  Physical component from baseline to week 24 | 0.90 (7.59) | 1.36 (3.74)
  Physical component from baseline to week 48 | 0.70 (5.98) | 2.41 (4.82)
  Physical component from week 24 to week 48 | -0.21 (6.80) | 1.05 (3.64)
  Mental component from baseline to week 24 | -3.08 (11.44) | -0.49 (2.02)
  Mental component from baseline to week 48 | -1.46 (7.74) | 0.49 (1.74)
  Mental component from week 24 to week 48 | 1.62 (11.46) | 0.98 (2.29)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 24; mITT LOCF. (Physical component score); Test type: Superiority; p = 0.8420, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 0.59, 95% CI 2-sided [-5.55 to 6.73] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 24; mITT LOCF. (Mental component score); Test type: Superiority; p = 0.6693, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.74, 95% CI 2-sided [-10.15 to 6.67] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 48; mITT LOCF. (Physical component score); Test type: Superiority; p = 0.5444, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.83, 95% CI 2-sided [-8.12 to 4.46] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 48; mITT LOCF. (Mental component score); Test type: Superiority; p = 0.5595, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.85, 95% CI 2-sided [-8.47 to 4.76] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Physical component score); Test type: Superiority; p = 0.4331, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.07, 95% CI 2-sided [-7.54 to 3.41] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; Week 24 to week 48; mITT LOCF. (Mental component score); Test type: Superiority; p = 0.6427, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -1.44, 95% CI 2-sided [-7.90 to 5.03] — [estimate comment as in outcome 10, analysis 1]

21. Secondary Outcome: Number of Participants With Adverse Event(s) and/or Serious Adverse Event(s) - Open-label Extension
Description: Number of participants with adverse event(s) and/or serious adverse event(s) reported from week 24 to week 48
Time Frame: from week 24 to week 48
Population: One subject was excluded from safety analysis (in the Tesofensine/Metoprolol -> Tesofensine/Metoprolol arm) since subject discontinued Tesomet treatment in Part 1 but continued in Part 2 without being dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 11 | 6
Participants
  Infections and infestations | 6 | 4
  Gastrointestinal disorders | 5 | 3
  Musculoskeletal and connective tissue disorders | 7 | 1
  Nervous system disorders | 3 | 4
  General disorders and administration site conditions | 4 | 0
  Psychiatric disorders | 2 | 2
  Cardiac disorders | 0 | 3
  Injury, poisoning and procedural complications | 1 | 1
  Vascular disorders | 0 | 2
  Blood and lymphatic system disorders | 1 | 0
  Investigations | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 1 | 0

22. Secondary Outcome: Blood Pressure (Change)
Description: Change in blood pressure from baseline to week 24, from baseline to week 48, and from week 24 to week 48. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
mmHg
  Change in Systolic BP from baseline to week 24 | 2.0 (13) | -4.2 (8)
  Change in Systolic BP from baseline to week 48 | 5.8 (14) | -9.7 (13)
  Change in Systolic BP from week 24 to wek 48 | 5.0 (11) | -5.5 (14)
  Change in Diastolic BP from baseline to week 24 | 2.8 (11) | -2.0 (11)
  Change in Diastolic BP from baseline to week 48 | 6.5 (12) | -1.0 (13)
  Change in Diastolic BP from week 24 to week 48 | 4.2 (9) | 1.0 (10)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 24; safety set LOCF. (Change in systolic blood pressure); Test type: Superiority; p = 0.3037, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 5.86, 95% CI 2-sided [-5.76 to 17.48] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 24; safety set LOCF. (Change in diastolic blood pressure); Test type: Superiority; p = 0.7912, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.15, 95% CI 2-sided [-7.85 to 10.16] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 48; safety set LOCF. (Change in systolic blood pressure); Test type: Superiority; p = 0.1773, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 10.29, 95% CI 2-sided [-5.25 to 25.83] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 48; safety set LOCF. (Change in diastolic blood pressure); Test type: Superiority; p = 0.7980, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.32, 95% CI 2-sided [-9.55 to 12.20] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From week 24 to week 48; safety set LOCF. (Change in systolic blood pressure); Test type: Superiority; p = 0.1580, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 7.77, 95% CI 2-sided [-3.40 to 18.94] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From week 24 to week 48; safety set LOCF. (Change in diastolic blood pressure); Test type: Superiority; p = 0.7021, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.64, 95% CI 2-sided [-7.36 to 10.64] — [estimate comment as in outcome 10, analysis 1]

23. Secondary Outcome: 24 Hours Blood Pressure
Description: Changes in 24 hours blood pressure from baseline to week 12 and baseline to week 24
Time Frame: from baseline to week 12 and baseline to week 24
Population: Number of participants analyzed:
  Tesofensine/Metoprolol - Baseline/Week 12/Week 24: 14/12/9 Placebo - Baseline/Week 12/Week24: 8/6/5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 12 | 6
mmHg
  Systolic BP mean change from baseline to week 12 | -8.0 (20) | 0.7 (14)
  Systolic BP mean change from baseline to week 24: number analyzed (Participants) | 9 | 5
  Systolic BP mean change from baseline to week 24 | 2.3 (20) | -8.4 (17)
  Diastolic BP mean change from baseline to week 12 | 0.2 (9) | 3.7 (8)
  Diastolic BP mean change from baseline to week 24: number analyzed (Participants) | 9 | 5
  Diastolic BP mean change from baseline to week 24 | 3.7 (8) | -2.8 (9)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; From baseline to week 24; mITT LOCF. (Change in systolic blood pressure mean); Test type: Superiority; p = 0.8728, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 1.50, 95% CI 2-sided [-18.17 to 21.18] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol vs Placebo; From baseline to week 24; mITT LOCF. (Change in diastolic blood pressure mean); Test type: Superiority; p = 0.5714, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.46, 95% CI 2-sided [-6.61 to 11.54] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol vs Placebo; From baseline to week 12; mITT LOCF. (Change in systolic blood pressure mean); Test type: Superiority; p = 0.2322, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -10.15, 95% CI 2-sided [-27.51 to 7.22] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Tesofensine/Metoprolol vs Placebo; From baseline to week 12; mITT LOCF. (Change in diastolic blood pressure mean); Test type: Superiority; p = 0.4321, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -3.46, 95% CI 2-sided [-12.61 to 5.68] — [estimate comment as in outcome 10, analysis 1]

24. Secondary Outcome: Plasma Trough Concentrations
Description: Plasma trough concentrations of tesofensine, metabolite NS2360 and metoprolol for the active arm (the first 24 weeks and then continuously up to week 48) and placebo arm (start of treatment at week 25 and then continuously up to week 48). mITT observed values.
Time Frame: baseline to week 48
Population: The Placebo -> Tesofensine/Metoprolol group did not start treatment before week 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 11 | 6
μg/L
  Tesofensine Week 12: number analyzed (Participants) | 11 | 0
  Tesofensine Week 12 | 12.03 (38.6) |
  Tesofensine Week 24: number analyzed (Participants) | 11 | 0
  Tesofensine Week 24 | 12.34 (55.4) |
  Tesofensine Week 36 | 11.01 (54.4) | 19.10 (56.1)
  Tesofensine Week 48 | 6.78 (394.7) | 15.11 (70.2)
  NS2360 metab. Week 12: number analyzed (Participants) | 11 | 0
  NS2360 metab. Week 12 | 3.39 (48.5) |
  NS2360 metab. Week 24: number analyzed (Participants) | 11 | 0
  NS2360 metab. Week 24 | 3.96 (71.9) |
  NS2360 metab. Week 36 | 3.39 (57.1) | 6.51 (56.3)
  NS2360 metab. Week 48 | 2.44 (157.3) | 6.02 (67.7)
  Metoprolol Week 12: number analyzed (Participants) | 11 | 0
  Metoprolol Week 12 | 10.83 (120.8) |
  Metoprolol Week 24: number analyzed (Participants) | 11 | 0
  Metoprolol Week 24 | 9.07 (281.4) |
  Metoprolol Week 36 | 8.97 (309.6) | 10.62 (206.0)
  Metoprolol Week 48 | 7.29 (156.9) | 7.30 (578.8)

25. Secondary Outcome: 48 Hours Heart Rate and QT Interval at Baseline, Week 12 and Week 24
Description: For Part 1, 48 hours HR and QT interval from week 12 to week 24 were not recorded in the database and analysis of changes not evaluated. Instead, abnormal findings over visits were summarized.
  Abnormal ECG findings detected in the three Tesomet treated subjects are:
  * QTc prolongation (466 ms)
  * Bradycardia (56 bpm)
  * QTc prolongation (460 ms) All were considered not clinically significant.
Time Frame: baseline, week 12 and week 24
Population: 21 sub. were assign. 22 randomization no.
  1 sub. was screen failure received 1 dose of Tesomet prior to being withdrawn at baseline. Sub. was re-screened and randomized as new sub. receiving PBO. As this sub. was assigned 2 randomization no., 1 under each arm, the sub. is summarized for both arms. The 2 randomization no. are considered as 2 sub.
  14 sub. were randomized to receive Tesomet and 8 sub. received PBO. 4 sub. (2 Tesomet, 2 PBO) terminated study before end of 24W DB period.
Measure: Count of Participants; unit: Participants
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 14 | 8
Participants
  ECG interretation baseline: Normal | 14 | 8
  ECG interretation baseline: Abnormal | 0 | 0
  ECG interretation at week 12: number analyzed (Participants) | 12 | 6
  ECG interretation at week 12: Normal | 9 | 6
  ECG interretation at week 12: Abnormal | 3 | 0
  ECG interretation at week 24: number analyzed (Participants) | 12 | 6
  ECG interretation at week 24: Normal | 11 | 6
  ECG interretation at week 24: Abnormal | 1 | 0
  48 hour heart rate at baseline: number analyzed (Participants) | 13 | 8
  48 hour heart rate at baseline: Normal | 13 | 8
  48 hour heart rate at baseline: Abnormal | 0 | 0
  48 hour heart rate at week 12: number analyzed (Participants) | 12 | 6
  48 hour heart rate at week 12: Normal | 10 | 6
  48 hour heart rate at week 12: Abnormal | 2 | 0
  48 hour heart rate at week 24: number analyzed (Participants) | 12 | 6
  48 hour heart rate at week 24: Normal | 12 | 6
  48 hour heart rate at week 24: Abnormal | 0 | 0

26. Secondary Outcome: Heart Rate (Change)
Description: Change in heart rate from baseline to week 24, from baseline to week 48, and from week 24 to week 48. mITT observed values.
Time Frame: from baseline to week 24, from baseline to week 48 and from week 24 to week 48
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
Number analyzed (Participants) | 12 | 6
bpm
  Change in Heart Rate from baseline to week 24 | -2.4 (11) | -7.0 (12)
  Change in Heart Rate from baseline to week 48 | 0.1 (7) | 0.7 (20)
  Change in Heart Rate from week 24 to week 48 | 4.2 (8) | 7.7 (10)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 24; safety set LOCF. (Change in heart rate); Test type: Superiority; p = 0.5551, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = 2.70, 95% CI 2-sided [-6.72 to 12.12] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From baseline to week 48; safety set LOCF. (Change in heart rate); Test type: Superiority; p = 0.7256, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -2.13, 95% CI 2-sided [-14.88 to 10.63] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tesofensine/Metoprolol -> Tesofensine/Metoprolol vs Placebo -> Tesofensine/Metoprolol; From week 24 to week 48; safety set LOCF. (Change in heart rate); Test type: Superiority; p = 0.4822, ANCOVA — P-value from an ANCOVA model with treatment as factor and baseline as covariate; LS Mean Difference = -3.29, 95% CI 2-sided [-13.05 to 6.48] — [estimate comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: Part 1 (double-blind part): From the first dose of double-blind study drug during Part 1 until the last dose during Part 1 (24 weeks duration). Part 2 (open-label extension part): From the first dose of open-label study drug during Part 2 until the last dose during Part 2 (24 weeks duration).
Description: Part 1: Safety Analysis Set included all subjects who took at least 1 dose of study drug (active substances or matching placebos).
  Part 2: Safety Analysis Set included all subjects who took at least 1 dose of study drug in the open-label extension (active substances or matching placebos); 1 subject continued in Part 2 without being dosed and was therefore excluded from the Safety Analysis Set.
Arm/Group | Tesofensine/Metoprolol | Placebo | Tesofensine/Metoprolol -> Tesofensine/Metoprolol | Placebo -> Tesofensine/Metoprolol
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/8 | 1/11 | 0/6
Other Adverse Events (participants affected / at risk) | 12/14 | 7/8 | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesofensine/Metoprolol (N=14) | Placebo (N=8) | Tesofensine/Metoprolol -> Tesofensine/Metoprolol (N=11) | Placebo -> Tesofensine/Metoprolol (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesofensine/Metoprolol (N=14) | Placebo (N=8) | Tesofensine/Metoprolol -> Tesofensine/Metoprolol (N=11) | Placebo -> Tesofensine/Metoprolol (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (5) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (9) | 3 (6) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 0 (0) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 7 (7) | 1 (1) | 2 (2) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Energy increased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03845075/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT03845075/SAP_001.pdf